CLINICAL TRIAL: NCT01862133
Title: Aspiring to Awesome- Patient Preference Privacy Selections in EMR
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Regenstrief Institute, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: CFDA# 93.719
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Results first posted 2015-03-23 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: Sexually Transmitted Diseases
Keywords: Electronic Health Record; Health Information Technology; Patient Privacy; Personal Health Information
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patient Preferences: Patients were eligible if they had visited their primary care physician at least twice in the previous 1 year and were fluent in English. Each patient subject used an online program to record their preferences what each of their providers can see. The electronic medical record (EMR) will then apply them to data displays.
- Primary Care Providers: All healthcare providers (physicians, nurses, and other clinic staff) were eligible to participate in this study. For those enrolled, display of patient data in the EMR was dictated by the patient subject's preferences for who should see what data.
  Interventions: Other: Patient preferences

INTERVENTIONS:
Other: Patient preferences — Software for recording patients' preferences for which providers see which parts of their EMRs, and EMR software for restricting access to data based on patients' preferences.
  Groups: Primary Care Providers

SUMMARY:
Health information technology, including health information exchange, offers the potential to improve care by providing an integrated view of relevant, integrated patient information from multiple health care providers practicing in multiple sites. However, realizing that potential can be difficult, particularly with respect sensitive information. Increasingly, patients, patient advocate groups, and even the National Coordinator for Health Information Technology are pushing for patients to have more granular control over specifically who can see what personal health information in their electronic health records.

This will be a demonstration project aimed at showing the initial feasibility a system allowing patient controls on their electronic health records. Because of the exploratory nature of the research, the investigators do not have specific hypotheses. The investigators hope that this demonstration and feasibility project will lead to more extensive prospective evaluations of patient control of access to their health records and other tools for enhancing patient control over access to their health records.

DETAILED DESCRIPTION:
In 2010, ONC launched a Challenge Grant program that called for proposals for "enabling enhanced query for patient care." Under this program, the Regenstrief Institute and Indiana University developed a Web-based program for patients' to express their preferences for who can access data in their electronic health records (EHR). It then applied these preferences by modifying an existing EHR viewer called Careweb® that is used by the Indiana Network for Patient Care and Eskenazi Health, an urban public health system in Indianapolis.

This study:

1. Produced a bioethical report on "points to consider" to inform electronic health record designers concerning giving patients granular control over access to their health data.
2. Interviewed patients to assess their desires for granular level of control over which personal health information should be shared, with whom, and for what purpose, and whether those preferences vary depending on the sensitivity of patients' health information.
3. Developed a Web-based patient-centered user interface that allows them to choose whether to provide or restrict access to their health information, focusing on who (health care providers and non-providers), what information (all, none, sensitive information only), and when (periods of time in their lives during which they desire restricting access to their health information) .
4. Reprogrammed the user interface of Careweb®, a data viewing system used by clinicians in Eskenazi Health, the third largest safety net health system in the U.S., and the Indiana Network for Patient Care, the oldest, largest, and most comprehensive health information exchange in the country. The reprogrammed viewer interface allows patients' preferences to control who sees what information in a patient's electronic health record.
5. Performed a demonstration study among 32 health care providers (9 physicians and 23 clinical staff) and 105 patients in an inner city primary care practice where patients recorded their preferences concerning who could access what information in their electronic health records, and then implemented those preferences during a 6-month real-world study in Eskenazi Health.

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* all adults 18 years or older who were fluent in English and had visited the study primary care clinic at least twice in the previous year

For Providers:

* all personnel of all types practicing in General Medicine Clinic, both Firms A and B, on the 4th floor of Wishard's Primary Care Center. For those physicians who agree to participate, attempted to recruit 10 patients who had visited their primary care physician at least twice in the previous 1 year.

Exclusion Criteria:

* will be lack of English fluency and inability to communicate due to physiologic or cognitive difficulties.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tierney, MD, Principal Investigator — Indiana University
Locations (1):
- Wishard Health Services, Primary Care Center, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Caine K, Tierney WM. Point and counterpoint: patient control of access to data in their electronic health records. J Gen Intern Med. 2015 Jan;30 Suppl 1(Suppl 1):S38-41. doi: 10.1007/s11606-014-3061-0. PMID 25480723
- [Background] Meslin EM, Schwartz PH. How bioethics principles can aid design of electronic health records to accommodate patient granular control. J Gen Intern Med. 2015 Jan;30 Suppl 1(Suppl 1):S3-6. doi: 10.1007/s11606-014-3062-z. PMID 25480724
- [Result] Leventhal JC, Cummins JA, Schwartz PH, Martin DK, Tierney WM. Designing a system for patients controlling providers' access to their electronic health records: organizational and technical challenges. J Gen Intern Med. 2015 Jan;30 Suppl 1(Suppl 1):S17-24. doi: 10.1007/s11606-014-3055-y. PMID 25480722
- [Result] Schwartz PH, Caine K, Alpert SA, Meslin EM, Carroll AE, Tierney WM. Patient preferences in controlling access to their electronic health records: a prospective cohort study in primary care. J Gen Intern Med. 2015 Jan;30 Suppl 1(Suppl 1):S25-30. doi: 10.1007/s11606-014-3054-z. PMID 25480721
- [Result] Tierney WM, Alpert SA, Byrket A, Caine K, Leventhal JC, Meslin EM, Schwartz PH. Provider responses to patients controlling access to their electronic health records: a prospective cohort study in primary care. J Gen Intern Med. 2015 Jan;30 Suppl 1(Suppl 1):S31-7. doi: 10.1007/s11606-014-3053-0. PMID 25480720
- [Result] Caine K, Kohn S, Lawrence C, Hanania R, Meslin EM, Tierney WM. Designing a patient-centered user interface for access decisions about EHR data: implications from patient interviews. J Gen Intern Med. 2015 Jan;30 Suppl 1(Suppl 1):S7-16. doi: 10.1007/s11606-014-3049-9. PMID 25480719

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 107 primary care clinic patients were enrolled and signed informed consent statements. 2 failed to complete the patient preference dialog and study questionnaire.
Groups:
- Patient Preferences: Patients were eligible if they had visited their primary care physician at least twice in the previous 1 year and were fluent in English. Each patient subject used an online program to record their preferences what each of their providers can see. The electronic medical record (EMR) will then apply them to data displays.
  141 adult primary care clinic patients were approached 38 refused to participate 107 were enrolled and signed informed consent statements 2 failed to complete the patient preference dialog and study questionnaire 105 completed the patient preference dialog and were included in the study 92 subjects returned to the clinic during the 6-month study
- Primary Care Providers: All healthcare providers (physicians, nurses, and other clinic staff) were eligible to participate in this study. For those enrolled, display of patient data in the EMR was dictated by the patient subject's preferences for who should see what data.
  Patient preferences: Software for recording patients' preferences for which providers see which parts of their EMRs, and EMR software for restricting access to data based on patients' preferences.
  * 11 physicians and 23 additional clinic staff (5 nurses, 4 clinical nurse assistants, 3 physicians' assistants, 2 nurse practitioners, and 9 medical assistance worked in the study primary care clinic at the time of the study
  * 2 physicians were excluded because their patients were mainly Spanish speaking
  * 1 physician verbally agreed to be in the study but never signed the informed consent statement
  * 8 physicians and all 23 of the other clinic staff were enrolled and signed informed consent statements and completed in the study
Period: Overall Study
Arm/Group | Patient Preferences | Primary Care Providers
Started | 105 | 31
Returned During 6 mo Study | 92 | 31
Completed | 105 (All 105 patients recorded preferences; 92 (88%) returned to the study clinic during the 6 mo. study) | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data collected from enrolled patients was limited to gender, race/ethnicity, age, and whether they had highly sensitive information (as defined in Methods) in their electronic health records. This information was obtained from patients' electronic medical records only.
Arm/Group | Patient Preferences
Number analyzed (Participants) | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Recording Preferences to Restrict Provider Access to Some or All Electronic Health Record (EHR) Data
Description: Patients had to restrict access to either all data or one of five categories of "sensitive" data (sexually transmitted infections, HIV/AIDS, sexual health and pregnancy, drug and alcohol use and abuse, and mental health information) to one or more of the study providers.
Time Frame: 6 month study
Population: All patients recorded their preferences and completed the questionnaire. 24 (77%) of the 31 providers completed the anonymous post-study questionnaire.
Measure: Number; unit: participants
Groups:
- Primary Care Providers: All healthcare providers (physicians, nurses, and other clinic staff) were eligible to participate in this study. For those enrolled, display of patient data in the EMR was dictated by the patient subject's preferences for who should see what data.
  Patient preferences: Software for recording patients' preferences for which providers see which parts of their EMRs, and EMR software for restricting access to data based on patients' preferences.
  * 11 physicians and 23 additional clinic staff (5 nurses, 4 clinical nurse assistants, 3 physicians' assistants, 2 nurse practitioners, and 9 medical assistance worked in the study primary care clinic at the time of the study
  * 2 physicians were excluded because their patients were mainly Spanish speaking
  * 1 physician verbally agreed to be in the study but never signed the informed consent statement
  * 8 physicians and all 23 of the other clinic staff were enrolled and signed informed consent statements and completed in the study
  * 24
Arm/Group | Patient Preferences | Primary Care Providers
Number analyzed (Participants) | 105 | 24
participants | 45 | 13

2. Primary Outcome: Providers' Opinion of Patients' Controlling EHR Access
Description: Percent of providers answering "Strongly Agree" or "Agree" to the following question on the post-study survey: "I think it is OK for patients to have control over who sees what information in their electronic health records."
Time Frame: 6 month study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: Patient complaints
Arm/Group | Patient Preferences | Primary Care Providers
Serious Adverse Events (participants affected / at risk) | 0/105 | 0/31
Other Adverse Events (participants affected / at risk) | 0/105 | 0/31

LIMITATIONS AND CAVEATS:
We could not separate the anonymous post-study provider survey results and comments by provider type because the numbers within the physicians and nurses were sufficiently small that anonymity could have been lost.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No